CLINICAL TRIAL: NCT03462979
Title: GlPs Improve Practice (GIP) at Home: Effects of Home Gluten Immunogenic Peptide Testing on Children With Celiac Disease
Brief Title: Effects of Home Gluten Immunogenic Peptide Testing on Children With Celiac Disease
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: covid-19 pandemic
Sponsor: Boston Children's Hospital (Other)
Collaborators: Glutenostics, LLC (Unknown)
Responsible Party: Principal Investigator, Jocelyn Silvester, Instructor, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P00024698
Record Dates: First submitted 2018-03-05; First posted 2018-03-13 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Celiac Disease; Gluten Sensitivity; Gluten Enteropathy; Gastrointestinal Disease; Digestive System Disease; Diet Modification; Intestinal Disease; Malabsorption Syndromes; Patient Compliance; Diagnostic Self Evaluation; Quality of Life
Keywords: Gluten-free diet; Urine; Stool; home testing
MeSH Terms: conditions — Celiac Disease; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases; Malabsorption Syndromes; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Results with home testing (Experimental): Participants in the open results arm will be provided with Gluten Detective home testing kits (immunochromatographic lateral flow tests) at week 8 of the study for immediate qualitative (yes/no) feedback about the presence of biomarkers of gluten in their stool and/or urine. During the period from week 8 to week 30, participants will be contacted a total of 6 times at random intervals to collect and test urine samples and complete a questionnaire.Additionally, participants will be given 4 stool test kits, with instructions that they may use these at times of their choosing and will report results and reasons for test use, if any. During this time participants will also keep a diary of suspected gluten exposures. All samples collected will be returned during the week 30 study visit.
  Interventions: Device: Immunochromatographic lateral flow test
- Blinded (sample collection only) (No Intervention): Participants in the blinded arms will not be given a test kit but will be given sample collection materials. During the period from week 8 to week 30 of the study, participants will be contacted a total of 6 times at random intervals, instructed to collect urine samples, and complete a questionnaire. Participants will also keep a diary of suspected gluten exposures. All samples collected will be returned during the week 30 study visit. After completion of sample collection, all participants will be unblinded and notified of the results once the samples have been processed.

INTERVENTIONS:
Device: Immunochromatographic lateral flow test — The immunochromatographic lateral flow test (Gluten Detective) is an at-home test that detects gluten immunogenic peptides excreted in stool or urine. This test can detect gluten exposures which occurred either during the last 24 hours (urine) or within up to a 7 day window (stool). Minimum intake amounts of gluten for successful detection using these test are 50mg (stool) to 500mg (urine)
  Other Names: Gluten Detective
  Arms: Open Results with home testing

SUMMARY:
This study aims to investigate how knowledge of gluten immunogenic peptide (GIP) levels in stool and urine affects subsequent adherence to a gluten-free diet. Half of the participants will receive results in real-time using a home device and the other half will store samples to be tested at the end of the 30 week study. Participants will also have a diet review with a dietitian at the beginning of the end of their study and be asked questions about their symptoms, gluten-free diet adherence and quality of life.

DETAILED DESCRIPTION:
Following a gluten-free diet is difficult. Eating small amounts of gluten may be common. Gluten may cause a wide range of symptoms, or no symptoms at all. Thus, there is not always a 'feedback loop' to alert to accidental gluten exposure. Nevertheless, these "silent" gluten exposures may interfere with recovery and healing of the intestine. New tools are available to test for fragments of gluten - Gluten Immunogenic Peptides (GIPs) in urine and stool.

The goal of this research study is to evaluate how knowledge of gluten-immunogenic peptide (GIP) levels in urine and stool affects subsequent adherence to a gluten-free diet. Participants will be children with celiac disease recruited at Boston Children's Hospital. All participants will undergo a diet assessment by a dietitian at the beginning and end of the study. At random intervals, participants will be prompted to collect their next urine sample and complete a survey related to symptoms and diet adherence. Half of the participants will store the sample to be tested later and the rest of the participants will be provided with devices to test their urine at home to receive immediate results. Participants in the home testing group will also be given a set of stool tests (x4) to use at their own discretion during the study period, and will report results and reasons for test use to the research team. GIP test results will be compared to other measures of celiac disease and gluten-free diet adherence, including antibody tests. These findings will help to determine how these new tools can be used to improve gluten-free diet adherence and symptoms and the effect on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 18 years at study entry
* Diagnosis of celiac disease based upon either

  1. Biopsy criteria i) Marsh 3 lesion and/or villous height:crypt depth ratio (Vh:Cd) < 3 with intraepithelial lymphocytosis; and ii) Elevated serum tTG IgA and/or EMA antibodies
  2. Serologic/genetic (ESPGHAN 2012) criteria i) Symptoms compatible with celiac disease; ii) Serum tTG IgA > 10 x upper limit of normal for assay; iii) EMA titre elevated on a separate sample; and iv) HLADQ genotype compatible with celiac disease.
* Adherence to a gluten-restricted diet (self-reported) for 6 months or more
* Attending a clinician assessment for celiac disease at Boston Children's Hospital

Exclusion Criteria:

* Unable to provide urine and/or stool sample or attend study visits
* English proficiency unsuitable for completion of surveys
* Anuria or oliguria
* Reliance upon commercial gluten-free formulas as primary source of nutrition
* Comorbid condition that in the opinion of the investigator would interfere with the subject's participation in the study or would confound the results of the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in frequency of gluten exposure in open results vs blinded groups following randomization. | Weeks 8 to 30
  Gluten exposure frequency is defined as the average per individual subject post-randomization percentage of samples collected between weeks 8 and 30 with detectable gluten immunogenic peptides using the qualitative assay (Gluten Detective)

SECONDARY OUTCOMES:
Difference in quantity of mean gluten exposure following randomization in blinded vs. open results groups | weeks 8 - 30
  Mean gluten exposure is defined as the average per individual subject post-randomization concentration of gluten immunogenic peptides detected using the quantitative assay
Celiac disease symptom score in blinded vs. open results group at the end of the study | Week 30
  Symptom score (using the Celiac Disease PedsRO or ObsRO as appropriate for age) at week 30
Change in symptom score in blinded vs. open results group | weeks 8 and 30
  Symptom score (using the Celiac Disease PedsRO or ObsRO as appropriate) and the change in symptom score between the end of the run-in period (week 8) and the end of the study period (week 30) will be calculated arithmetically.
Change in celiac disease specific quality of life as measured by Celiac Disease DUX (CDDUX) in blinded vs. open results groups | weeks 8 and 30
  The CDDUX is a disease specific quality of life instrument for children with celiac disease.
Change in pediatric health related quality of life as measured by PedsQL 4.0 generic core scale in blinded vs. open results groups | weeks 8 and 30
  The PedsQL 4.0 Generic Core is a validated pediatric general quality of life measure that is caregiver reported for younger children and both child and caregiver reported for older children. The score is scaled from 0 (lowest) to 100 (highest) with higher scores corresponding to better health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn A Silvester, MD PhD, Principal Investigator — Boston Children's Hospital, Beth Israel Deaconess Medical Center
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreno ML, Cebolla A, Munoz-Suano A, Carrillo-Carrion C, Comino I, Pizarro A, Leon F, Rodriguez-Herrera A, Sousa C. Detection of gluten immunogenic peptides in the urine of patients with coeliac disease reveals transgressions in the gluten-free diet and incomplete mucosal healing. Gut. 2017 Feb;66(2):250-257. doi: 10.1136/gutjnl-2015-310148. Epub 2015 Nov 25. PMID 26608460
- [Background] Comino I, Real A, Vivas S, Siglez MA, Caminero A, Nistal E, Casqueiro J, Rodriguez-Herrera A, Cebolla A, Sousa C. Monitoring of gluten-free diet compliance in celiac patients by assessment of gliadin 33-mer equivalent epitopes in feces. Am J Clin Nutr. 2012 Mar;95(3):670-7. doi: 10.3945/ajcn.111.026708. Epub 2012 Jan 18. PMID 22258271
- [Background] Comino I, Fernandez-Banares F, Esteve M, Ortigosa L, Castillejo G, Fambuena B, Ribes-Koninckx C, Sierra C, Rodriguez-Herrera A, Salazar JC, Caunedo A, Marugan-Miguelsanz JM, Garrote JA, Vivas S, Lo Iacono O, Nunez A, Vaquero L, Vegas AM, Crespo L, Fernandez-Salazar L, Arranz E, Jimenez-Garcia VA, Antonio Montes-Cano M, Espin B, Galera A, Valverde J, Giron FJ, Bolonio M, Millan A, Cerezo FM, Guajardo C, Alberto JR, Rosinach M, Segura V, Leon F, Marinich J, Munoz-Suano A, Romero-Gomez M, Cebolla A, Sousa C. Fecal Gluten Peptides Reveal Limitations of Serological Tests and Food Questionnaires for Monitoring Gluten-Free Diet in Celiac Disease Patients. Am J Gastroenterol. 2016 Oct;111(10):1456-1465. doi: 10.1038/ajg.2016.439. Epub 2016 Sep 20. PMID 27644734
- [Background] Shan L, Molberg O, Parrot I, Hausch F, Filiz F, Gray GM, Sollid LM, Khosla C. Structural basis for gluten intolerance in celiac sprue. Science. 2002 Sep 27;297(5590):2275-9. doi: 10.1126/science.1074129. PMID 12351792
- [Background] Moron B, Bethune MT, Comino I, Manyani H, Ferragud M, Lopez MC, Cebolla A, Khosla C, Sousa C. Toward the assessment of food toxicity for celiac patients: characterization of monoclonal antibodies to a main immunogenic gluten peptide. PLoS One. 2008 May 28;3(5):e2294. doi: 10.1371/journal.pone.0002294. PMID 18509534
- [Background] van Doorn RK, Winkler LM, Zwinderman KH, Mearin ML, Koopman HM. CDDUX: a disease-specific health-related quality-of-life questionnaire for children with celiac disease. J Pediatr Gastroenterol Nutr. 2008 Aug;47(2):147-52. doi: 10.1097/MPG.0b013e31815ef87d. PMID 18664865
- [Background] Varni JW, Burwinkle TM, Seid M. The PedsQL 4.0 as a school population health measure: feasibility, reliability, and validity. Qual Life Res. 2006 Mar;15(2):203-15. doi: 10.1007/s11136-005-1388-z. PMID 16468077
- [Background] Silvester JA, Graff LA, Rigaux L, Walker JR, Duerksen DR. Symptomatic suspected gluten exposure is common among patients with coeliac disease on a gluten-free diet. Aliment Pharmacol Ther. 2016 Sep;44(6):612-9. doi: 10.1111/apt.13725. Epub 2016 Jul 22. PMID 27443825
- [Background] Lebwohl B, Sanders DS, Green PHR. Coeliac disease. Lancet. 2018 Jan 6;391(10115):70-81. doi: 10.1016/S0140-6736(17)31796-8. Epub 2017 Jul 28. PMID 28760445
- [Background] Ludvigsson JF, Ciacci C, Green PH, Kaukinen K, Korponay-Szabo IR, Kurppa K, Murray JA, Lundin KEA, Maki MJ, Popp A, Reilly NR, Rodriguez-Herrera A, Sanders DS, Schuppan D, Sleet S, Taavela J, Voorhees K, Walker MM, Leffler DA. Outcome measures in coeliac disease trials: the Tampere recommendations. Gut. 2018 Aug;67(8):1410-1424. doi: 10.1136/gutjnl-2017-314853. Epub 2018 Feb 13. PMID 29440464

DOCUMENTS (2):
  • Study Protocol (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/79/NCT03462979/Prot_004.pdf
  • Informed Consent Form (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT03462979/ICF_006.pdf